CLINICAL TRIAL: NCT01581151
Title: Dexamethasone Implant With Rescue Ranibizumab for Treating Macular Edema Secondary to Retinal Vein Occlusion
Brief Title: Ozurdex With Rescue Lucentis for Treating Macular Edema Secondary to Retinal Vein Occlusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brian Burke, MPH (Other)
Responsible Party: Sponsor-Investigator, Brian Burke, MPH, Investigator, Wills Eye
Organization: Wills Eye (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WE IRB# 11-122
Record Dates: First submitted 2012-04-17; First posted 2012-04-20 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Retinal Vein Occlusion
Keywords: retinal vein occlusion; ozurdex; lucentis; BCVA; foveal thickness
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Dexamethasone; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monthly Ranibizumab (Active Comparator): • Patients will receive a ranibizumab intravitreal injection on day 0. During each other visit, patients will receive a ranibizumab intravitreal injection. The protocol will use the term "monthly" to represent a 30 day interval between treatments.
  Interventions: Drug: Monthly Ranibizumab
- Dexamethasone intravitreal implant (Experimental): * Patients will receive a dexamethasone intravitreal implant injection at day 0.
  * During monthly visits 1,2,3, and 5, patients will receive a ranibizumab intravitreal injection if the macula SD-OCT during that visit shows mean central foveal thickness ≥ 250 μm or the best-corrected visual acuity is 20/40 or worse. The injection procedure is described in the next section.
  * During monthly visit 4, patients will receive a dexamethasone intravitreal implant injection if the macula SD-OCT during that visit shows mean central foveal thickness ≥ 250 μm or the best-corrected visual acuity is 20/40 or worse.
  Interventions: Drug: Dexamethasone intravitreal implant

INTERVENTIONS:
Drug: Dexamethasone intravitreal implant — Patients will receive a Dexamethasone implant and ranibizumab, as needed. A comparison will be made between ranibizumab and Dexamethasone implant with rescue ranibizumab.
  Other Names: Ozurdex - Allergan; Ranibizumab - Genentech
  Arms: Dexamethasone intravitreal implant
Drug: Monthly Ranibizumab — 30 days between treatments
  Other Names: Ranibizumab
  Arms: Monthly Ranibizumab

SUMMARY:
This study seeks to compare dexamethasone implant with rescue intravitreal ranibizumab to monthly intravitreal ranibizumab for the treatment of macular edema secondary to branch or central retinal vein occlusion. This is based on the null hypothesis that dexamethasone implant with rescue ranibizumab has inferior best corrected visual acuity at six months compared to monthly ranibizumab alone.

DETAILED DESCRIPTION:
Dexamethasone intravitreal implant (DEX implant; OZURDEX, Allergan, Inc., Irvine, CA) and Ranibizumab (Lucentis, Genentech, Inc., South San Francisco, CA) as needed group:

* Patients will receive a dexamethasone intravitreal implant injection at day 0. Injection procedure will be identical to those previously described.8,19,20 Topical tetracaine drops will be given, a lid speculum inserted, and then 5% povidone iodine drops will be given. After subconjunctival injection of 2% lidocaine, the 0.7mg DEX implant will be inserted through the pars plana using a customized, single use, 22-gauge applicator. Patients will be treated with topical ophthalmic antibiotics four times daily for three days after the procedure.
* During monthly visits 1,2,3, and 5, patients will receive a ranibizumab intravitreal injection if the macula SD-OCT during that visit shows mean central foveal thickness ≥ 250 μm or the best-corrected visual acuity is 20/40 or worse. The injection procedure is described in the next section.
* During monthly visit 4, patients will receive a dexamethasone intravitreal implant injection if the macula SD-OCT during that visit shows mean central foveal thickness ≥ 250 μm or the best-corrected visual acuity is 20/40 or worse.

Monthly Ranibizumab (Lucentis, Genentech, Inc., South San Francisco, CA) group:

* Patients will receive a ranibizumab intravitreal injection on day 0. During each other visit, patients will receive a ranibizumab intravitreal injection. The protocol will use the term "monthly" to represent a 30 day interval between treatments. The minimal interval between treatments may be 25 days.
* Injection procedures will be identical to those previously described.8,19,20 Topical tetracaine drops will be given, a lid speculum inserted, and then 5% povidone iodine drops will be given. After subconjunctival injection of 2% lidocaine, a 30-gauge needle will be inserted through the pars plana, and 0.5 mg (0.05mL) of drug injected.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* 18 to 90 year-old men or women
* Women must be postmenopausal for at least 12 months before study enrollment, or surgically sterile. Potential child bearing women must have a negative serum pregnancy test within 14 days prior to the first treatment and practice effective contraception during and at least 120 days following the last dose of injection.
* Patient of the Wills Eye Institute Retina service, including all Mid-Atlantic Retina offices.
* Healthy enough to participate in the study.
* Willing and able to consent to participation in the study.
* Retinal vein occlusion:
* Must be diagnosed within two weeks of onset of symptoms
* Best Corrected Visual Acuity (BCVA) on initial presentation between 20/40 and 20/320
* No contraindications to intravitreal injection of dexamethasone implant or ranibizumab
* Central foveal thickness greater than 250 m on Spectral Domain-OCT

Exclusion Criteria:

* Unknown duration of symptoms prior to diagnosis.
* Patients with any history of prior intravitreal dexamethasone or anti-VEGF or grid laser.
* Patients with diabetic retinopathy.
* Patients with age-related macular degeneration.
* Patients with an optic neuropathy.
* Patients with a retinal detachment or history of retinal detachment.
* Patients with a significant epiretinal membrane.
* Patients with a history of choroidal neovascularization.
* Patients with glaucoma with visual field loss documented on a Humphrey Visual Field test or ocular hypertension requiring more than 2 medications to control IOP in the study eye.
* Patients with a clinically significant media opacity.
* Patients using or anticipating using systemic steroids.
* Patients with any uncontrolled systemic disease.
* Patients with aphakia or anterior-chamber intraocular lens.
* Patients with active neovascularization of the iris, disc, or retina.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | 6 months
  • Primary outcome: Mean change from baseline in best corrected visual acuity score

SECONDARY OUTCOMES:
Foveal Thickness | 6 months
  * Mean absolute change from baseline in central foveal thickness,
  * Proportion of subjects with a central foveal thickness 250m
  * Mean change in fluid and central foveal thickness on OCT Time Frame
  * Proportion of subjects who gain at least 15 letters in BCVA score
  * Proportion of subjects who lose fewer than 15 letters in BCVA score
  * The incidence of ocular and systemic adverse events
  * Mean change from baseline in the NEI VFQ 25 near activities
  * Mean change from baseline in the NEI VFQ 25 distance activities

CONTACTS AND LOCATIONS:
Locations (1):
- Wills Eye Retina Service, Philadelphia, Pennsylvania, United States